CLINICAL TRIAL: NCT02437643
Title: An Enhanced Protein (Dairy) Weight Loss Intervention for Dynapenic Obesity: Impact on Muscle Quality and Composition
Acronym: DDYNAMO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Dairy Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pro00057509
Record Dates: First submitted 2015-05-05; First posted 2015-05-07 (Estimated); Last update posted 2018-11-07 (Actual); Status verified 2018-11

CONDITIONS: Dynapenia; Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- WL-LoEX (Placebo Comparator): 10% Weight loss diet plus low intensity exercise (protein ~0.8g/kg). Participants will be provided one serving of dairy protein daily.
  Interventions: Behavioral: Weight Loss; Dietary Supplement: Dairy Protein; Behavioral: Low intensity exercise
- Pro-WL-LoEX (Active Comparator): Protein-enhanced 10% Weight loss diet plus low intensity exercise (protein ~1.2 g/kg with > 30g per meal and >60% as dairy). Participants will be provided at least 8 servings of dairy protein daily.
  Interventions: Behavioral: Weight Loss; Dietary Supplement: Dairy Protein; Behavioral: Low intensity exercise

INTERVENTIONS:
Behavioral: Weight Loss — Participants will be prescribed hypo-caloric diet prescription.
Dietary Supplement: Dairy Protein — Participants will be provided dairy products: WL-LoEx will be provided 1 dairy serving per day and Pro-WL-LoEx will be provided 8 dairy servings per day.
Behavioral: Low intensity exercise — Participants in both groups will participate in chair exercises 3 times a week.

SUMMARY:
The purpose of the trial is to assess the effects of combining regular, generous intakes of high quality protein (primarily from dairy and other animal source proteins) with calorie restriction and low-intensity exercise on muscle quality and muscle adipose infiltration (along with bone mineral density [BMD] and a number of secondary outcomes) in frail, obese, older adults participating in a 6 month intervention. The investigators will compare these effects to those of a traditional control regimen of calorie restriction and low-intensity exercise over the same duration.

DETAILED DESCRIPTION:
Obese older adults (≥60 yrs) with moderate functional impairment will be randomized to 1 of 2 study arms. Outcomes to be measured at 0, 3 and 6 months are as follows: Primary outcomes- (1) Muscle Quality (MQ): muscle power (time to perform ten chair rises, height of the chair, leg length, body mass, and acceleration of gravity) in relation to muscle mass (CT-scan) and (2) Muscle adipose infiltration (MAI) (CT-scan). Secondary outcomes- Bone Mineral Density (BMD; DXA scan) physical function (Short Physical Performance Battery (SPPB); 6 minute walk; 8-foot up and go; and 30 second chair stands; handgrip strength; body weight; fat mass; waist circumference; activity (accelerometers); mental health (sleep, depression, quality of life); and feasibility factors (adherence, protein intake, nutrition adequacy). BMD will only be accessed at 0 and 6 months.

Study Arms:

* Weight loss plus low-intensity exercise intervention (WL-LoEX; n = 35): Subjects follow a calorie-reduction diet for a weight loss of ≥10%, protein~0.8g/g/d. Subjects will also participate in three 30-minute low-intensity exercise sessions weekly. One serving of dairy protein/day will be provided to WL-LoEX participants.
* High protein weight loss plus low-intensity exercise intervention (PRO-WL-LoEX; n = 35): Subjects follow a calorie-reduction diet for a weight loss of ≥10%, with a high proportion of high quality protein at each meal. Intakes of > 30g of protein will be achieved three times a day by subjects in this group, with all or predominantly all from animal sources (high quality) and 60-70% of animal protein from dairy foods that will be provided. Subjects will also participate in three 30-minute low-intensity exercise sessions weekly.

ELIGIBILITY:
Inclusion Criteria:

* BMI >30;
* SPPB score of ≥4 to <10;
* GFR <45 mL/min

Exclusion Criteria:

* Body weight >495 lbs. (BodPod limits);
* estimated glomerular filtration rates (eGFR) less than 45 mL/min;
* symptomatic cardiac disease;
* receiving chemotherapy;
* hemophilia;
* presence of unstable or symptomatic life-threatening illness;
* neurological disease or disorder causing functional impairments;
* inability to walk,
* dementia;
* prescription weight loss medications;
* use of monamine oxidase inhibitors (MAOIs); or
* primary medical provider advises against participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2018-10-15 (Actual); Study Completion 2018-10-15 (Actual)

PRIMARY OUTCOMES:
Change in muscle quality | baseline, 3 months, 6 months
  composite score of time to perform ten chair rises, height of the chair, leg length, body mass, and acceleration of gravity in relation to muscle mass
Change in muscle adipose infiltration | baseline, 3 months, 6 months
  CT-scan

SECONDARY OUTCOMES:
Change in Physical Function | baseline, 3 months, 6 months
  short physical performance battery score
Change in Body weight | baseline, 3 months, 6 months
  change in weight
Change in lean Body Mass | baseline, 3 months, 6 months
  BodPod
Change in lean Body Mass | baseline, 3 months, 6 months
  DEXA
Change in fat mass | baseline, 3 months, 6 months
  BodPod
Change in fat mass | baseline, 3 months, 6 months
  DEXA
Change in 6-minute walk time | baseline, 3 months, 6 months
  6-minute walk
Change in 8-foot up and go time | baseline, 3 months, 6 months
  time it takes to complete 8-foot up and go
Change in 30 second chair stands | baseline, 3 months, 6 months
  number of chair stands done in 30 seconds
Change in dietary protein intake | baseline, 3 months, 6 months
  3-day food record
Change in calorie intake | baseline, 3 months, 6 months
  3-day food record
Change in Bone Mineral Density | Baseline and 6-months
  DEXA
Change in sleep | baseline, 3 months, 6 months
  Pittsburgh sleep quality index
Change in depression | baseline, 3 months, 6 months
  Center for Epidemiologic Studies Depression Scale
Change in hand grip strength | baseline, 3 months, 6 months
  Jamar Hand Dynamometer
Change in physical activity | baseline, 3 months, 6 months
  Community Health Activities Model Program for Seniors (CHAMPS)
Change in physical activity | Baseline, 3 months, 6 months
  Actigraph - accelerometer
Change in quality of life | Baseline, 3 months, 6 months
  SF-36

CONTACTS AND LOCATIONS:
Overall Officials: Connie Bales, PhD, RD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Miller MG, Porter Starr KN, Rincker J, Orenduff MC, McDonald SR, Pieper CF, Fruik AR, Lyles KW, Bales CW. Rationale and Design for a Higher (Dairy) Protein Weight Loss Intervention That Promotes Muscle Quality and Bone Health in Older Adults with Obesity: A Randomized, Controlled Pilot Study. J Nutr Gerontol Geriatr. 2021 Apr-Jun;40(2-3):150-170. doi: 10.1080/21551197.2021.1896615. Epub 2021 Mar 13. PMID 33719918